CLINICAL TRIAL: NCT00005772
Title: Randomized Controlled Trial of Hypothermia for Hypoxic-Ischemic Encephalopathy in Term Infants
Brief Title: Whole-Body Cooling for Birth Asphyxia in Term Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0021; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD040461 (NIH); U10HD040492 (NIH); U10HD040498 (NIH); U10HD040521 (NIH); U10HD040689 (NIH); M01RR000030 (NIH); M01RR000039 (NIH); M01RR000044 (NIH); M01RR000070 (NIH); M01RR000080 (NIH); M01RR000633 (NIH); M01RR000750 (NIH); M01RR006022 (NIH); M01RR007122 (NIH); M01RR008084 (NIH); M01RR016587 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Hypoxia-Ischemia, Brain
Keywords: NICHD Neonatal Research Network; Hypoxic-ischemic encephalopathy (HIE); Hypothermia; Neonatal depression; Perinatal asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia (Experimental): Induced Whole-body hypothermia (with a target esophageal temperature of 33.5°C) for 96 hours
  Interventions: Device: Induced hypothermia
- Normothermic (Placebo Comparator): Placebo: Normothermic control group (with esophageal temperature at or near 37.0°C) for 96 hours
  Interventions: Device: Control

INTERVENTIONS:
Device: Induced hypothermia — Whole-body cooling using the Blanketrol II or III Units in the Automatic Control Mode with a YSI 400 series temperature probe placed in the distal esophagus over a 96-hour period
  Arms: Hypothermia
Device: Control — Control group: standard care
  Arms: Normothermic

SUMMARY:
This large multicenter trial tested whether cerebral cooling initiated within 6 hours of birth and continued for 72 hours would reduce the risk of death and moderate to severe neurodevelopmental injury at 18-22 months corrected age. Infants at least 36 weeks gestation with an abnormal blood gas within 1 hour of birth, or a history of an acute perinatal event and a 10-min Apgar score <5, or continued need for ventilation were screened. Following a neurological exam, those with moderate to severe encephalopathy were randomized to a 72-hour period of total body cooling (cooling blanket, followed by slow re-warming). The study was conducted in two phases: Phase I (20 infants) were examined for the safety of an esophageal temperature of 34-35 C; Phase II (main trial, 200 infants) were evaluated for the safety and efficacy of an esophageal temperature of 33-34 C. Cardio-respiratory, electroencephalograms (EEGs), renal, metabolic, and hematologic status, and esophageal and abdominal skin temperature were monitored during the 72 hours of intervention. Surviving children were given neurodevelopmental examinations at 18-22 months corrected age and again at school age (6-7 years of age).

DETAILED DESCRIPTION:
Perinatal cerebral hypoxia-ischemia injury is an important cause of death and neurodevelopmental disability. Data from animal models suggest that brain cooling immediately after injury is neuroprotective. Experience with total body cooling during surgery, accidental near drownings, and one Phase I trial of term infants suggest that it is effective and safe in children.

This large multicenter trial tested whether cerebral cooling initiated within 6 hours of birth and continued for 72 hours would reduce the risk of death and moderate to severe neurodevelopmental injury at 18-22 months corrected age. Infants at least 36 weeks gestation with an abnormal blood gas within 1 hour of birth, or a history of an acute perinatal event and a 10-min Apgar score <5, or continued need for ventilation were screened. Following a neurological exam, those with moderate to severe encephalopathy were randomized to a 72-hour period of total body cooling (cooling blanket, followed by slow re-warming). The study was conducted in two phases: Phase I (20 infants) were examined for the safety of an esophageal temperature of 34-35 C; Phase II (main trial, 200 infants) were evaluated for the safety and efficacy of an esophageal temperature of 33-34 C. Cardio-respiratory, electroencephalograms (EEGs), renal, metabolic, and hematologic status, and esophageal and abdominal skin temperature were monitored during the 72 hours of intervention.

Neurodevelopmental outcome was assessed at 18-22 mos of age by masked certified examiners. The outcome at 18-22 months showed that whole-body cooling reduces the risk of death or moderate to severe disability in infants with hypoxic ischemic encephalopathy.

Surviving infants were assessed at 6-7 years (school age).

ELIGIBILITY:
Inclusion Criteria:

* At least 36 weeks gestation
* Any blood gas (cord, postnatal) done within the first 60 minutes had a pH less than or equal to 7.0
* Any blood gas (cord postnatal) done within the first 60 minutes had a base deficit greater than or equal to 16 mEq/L
* All infants must have seizures or signs of moderate to severe encephalopathy before randomization

Exclusion Criteria:

* Inability to randomize by 6 hours of age
* Presence of known chromosomal anomaly or major congenital anomaly
* Severe intrauterine growth restriction (weight less than 1800g)
* All blood gases done within the first 60 minutes had a pH less than 7.15 and a base deficit less than 10 mEq/L
* Infants in extremis for whom no additional intensive therapy will be offered by attending neonatologist
* Parents refuse consent
* Attending neonatologist refuses consent

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 1999-10; Primary Completion 2003-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Death or moderate or severe disability | 18-22 months corrected age

SECONDARY OUTCOMES:
Length of hospital stay | Until discharge
Frequency of multi-organ dysfunction | Until discharge
Withdrawal of support | Until discharge
Post-neonatal deaths | 18-22 months corrected age
Multiple disability | 18-22 months corrected age
Seizure disorders | 18-22 months corrected age
Rehospitalizations | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Seetha Shankaran, MD, Principal Investigator — Wayne State University; Abbot R. Laptook, MD, Principal Investigator — Brown University, Womens and Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Study Director — Stanford University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Shahnaz Duara, MD, Principal Investigator — University of Miami; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; T. Michael O'Shea, MD, Principal Investigator — Wake Forest University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Harvard University, Cambridge, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Background] Shankaran S, Laptook A. Challenge of conducting trials of neuroprotection in the asphyxiated term infant. Semin Perinatol. 2003 Aug;27(4):320-32. doi: 10.1016/s0146-0005(03)00047-8. PMID 14510323
- [Background] Shankaran S. Neonatal encephalopathy: treatment with hypothermia. J Neurotrauma. 2009 Mar;26(3):437-43. doi: 10.1089/neu.2008.0678. PMID 19281415
- [Background] Higgins RD, Shankaran S. Hypothermia for hypoxic ischemic encephalopathy in infants > or =36 weeks. Early Hum Dev. 2009 Oct;85(10 Suppl):S49-52. doi: 10.1016/j.earlhumdev.2009.08.015. Epub 2009 Sep 17. PMID 19762176
- [Result] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Result] Shankaran S, Laptook A, Wright LL, Ehrenkranz RA, Donovan EF, Fanaroff AA, Stark AR, Tyson JE, Poole K, Carlo WA, Lemons JA, Oh W, Stoll BJ, Papile LA, Bauer CR, Stevenson DK, Korones SB, McDonald S. Whole-body hypothermia for neonatal encephalopathy: animal observations as a basis for a randomized, controlled pilot study in term infants. Pediatrics. 2002 Aug;110(2 Pt 1):377-85. doi: 10.1542/peds.110.2.377. PMID 12165594
- [Result] Ambalavanan N, Carlo WA, Shankaran S, Bann CM, Emrich SL, Higgins RD, Tyson JE, O'Shea TM, Laptook AR, Ehrenkranz RA, Donovan EF, Walsh MC, Goldberg RN, Das A; National Institute of Child Health and Human Development Neonatal Research Network. Predicting outcomes of neonates diagnosed with hypoxemic-ischemic encephalopathy. Pediatrics. 2006 Nov;118(5):2084-93. doi: 10.1542/peds.2006-1591. PMID 17079582
- [Result] Oh W, Perritt R, Shankaran S, Merritts M, Donovan EF, Ehrenkranz RA, O'Shea TM, Tyson JE, Laptook AR, Das A, Higgins RD. Association between urinary lactate to creatinine ratio and neurodevelopmental outcome in term infants with hypoxic-ischemic encephalopathy. J Pediatr. 2008 Sep;153(3):375-8. doi: 10.1016/j.jpeds.2008.03.041. Epub 2008 May 9. PMID 18534246
- [Result] Mietzsch U, Parikh NA, Williams AL, Shankaran S, Lasky RE. Effects of hypoxic-ischemic encephalopathy and whole-body hypothermia on neonatal auditory function: a pilot study. Am J Perinatol. 2008 Aug;25(7):435-41. doi: 10.1055/s-0028-1083842. Epub 2008 Aug 21. PMID 18720323
- [Result] Laptook A, Tyson J, Shankaran S, McDonald S, Ehrenkranz R, Fanaroff A, Donovan E, Goldberg R, O'Shea TM, Higgins RD, Poole WK; National Institute of Child Health and Human Development Neonatal Research Network. Elevated temperature after hypoxic-ischemic encephalopathy: risk factor for adverse outcomes. Pediatrics. 2008 Sep;122(3):491-9. doi: 10.1542/peds.2007-1673. PMID 18762517
- [Result] Shankaran S, Pappas A, Laptook AR, McDonald SA, Ehrenkranz RA, Tyson JE, Walsh M, Goldberg RN, Higgins RD, Das A; NICHD Neonatal Research Network. Outcomes of safety and effectiveness in a multicenter randomized, controlled trial of whole-body hypothermia for neonatal hypoxic-ischemic encephalopathy. Pediatrics. 2008 Oct;122(4):e791-8. doi: 10.1542/peds.2008-0456. PMID 18829776
- [Result] Parikh NA, Lasky RE, Garza CN, Bonfante-Mejia E, Shankaran S, Tyson JE. Volumetric and anatomical MRI for hypoxic-ischemic encephalopathy: relationship to hypothermia therapy and neurosensory impairments. J Perinatol. 2009 Feb;29(2):143-9. doi: 10.1038/jp.2008.184. Epub 2008 Nov 20. PMID 19020525
- [Result] Lasky RE, Parikh NA, Williams AL, Padhye NS, Shankaran S. Changes in the PQRST intervals and heart rate variability associated with rewarming in two newborns undergoing hypothermia therapy. Neonatology. 2009;96(2):93-5. doi: 10.1159/000205385. Epub 2009 Mar 2. PMID 19252411
- [Result] Laptook AR, Shankaran S, Ambalavanan N, Carlo WA, McDonald SA, Higgins RD, Das A; Hypothermia Subcommittee of the NICHD Neonatal Research Network. Outcome of term infants using apgar scores at 10 minutes following hypoxic-ischemic encephalopathy. Pediatrics. 2009 Dec;124(6):1619-26. doi: 10.1542/peds.2009-0934. PMID 19948631
- [Result] Kwon JM, Guillet R, Shankaran S, Laptook AR, McDonald SA, Ehrenkranz RA, Tyson JE, O'Shea TM, Goldberg RN, Donovan EF, Fanaroff AA, Poole WK, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Clinical seizures in neonatal hypoxic-ischemic encephalopathy have no independent impact on neurodevelopmental outcome: secondary analyses of data from the neonatal research network hypothermia trial. J Child Neurol. 2011 Mar;26(3):322-8. doi: 10.1177/0883073810380915. Epub 2010 Oct 4. PMID 20921569
- [Result] MacKay VL, Welch SK, Insley MY, Manney TR, Holly J, Saari GC, Parker ML. The Saccharomyces cerevisiae BAR1 gene encodes an exported protein with homology to pepsin. Proc Natl Acad Sci U S A. 1988 Jan;85(1):55-9. doi: 10.1073/pnas.85.1.55. PMID 3124102
- [Derived] Bonifacio SL, Chalak LF, Van Meurs KP, Laptook AR, Shankaran S. Neuroprotection for hypoxic-ischemic encephalopathy: Contributions from the neonatal research network. Semin Perinatol. 2022 Nov;46(7):151639. doi: 10.1016/j.semperi.2022.151639. Epub 2022 Jun 10. PMID 35835616
- [Derived] Pappas A, Shankaran S, McDonald SA, Carlo WA, Laptook AR, Tyson JE, Das A, Skogstrand K, Hougaard DM, Higgins RD. Blood Biomarkers and 6- to 7-Year Childhood Outcomes Following Neonatal Encephalopathy. Am J Perinatol. 2022 May;39(7):732-749. doi: 10.1055/s-0040-1717072. Epub 2020 Oct 10. PMID 33038899
- [Derived] Shankaran S, Laptook AR, McDonald SA, Hintz SR, Barnes PD, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health, and Human Development Neonatal Research Network. Acute Perinatal Sentinel Events, Neonatal Brain Injury Pattern, and Outcome of Infants Undergoing a Trial of Hypothermia for Neonatal Hypoxic-Ischemic Encephalopathy. J Pediatr. 2017 Jan;180:275-278.e2. doi: 10.1016/j.jpeds.2016.09.026. Epub 2016 Oct 21. PMID 27776752
- [Derived] Shankaran S, McDonald SA, Laptook AR, Hintz SR, Barnes PD, Das A, Pappas A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal Magnetic Resonance Imaging Pattern of Brain Injury as a Biomarker of Childhood Outcomes following a Trial of Hypothermia for Neonatal Hypoxic-Ischemic Encephalopathy. J Pediatr. 2015 Nov;167(5):987-93.e3. doi: 10.1016/j.jpeds.2015.08.013. Epub 2015 Sep 16. PMID 26387012
- [Derived] Vohr BR, Stephens BE, McDonald SA, Ehrenkranz RA, Laptook AR, Pappas A, Hintz SR, Shankaran S, Higgins RD, Das A; Extended Hypothermia Follow-up Subcommittee of the NICHD Neonatal Research Network. Cerebral palsy and growth failure at 6 to 7 years. Pediatrics. 2013 Oct;132(4):e905-14. doi: 10.1542/peds.2012-3915. Epub 2013 Sep 9. PMID 24019415
- [Derived] Shankaran S, Pappas A, McDonald SA, Vohr BR, Hintz SR, Yolton K, Gustafson KE, Leach TM, Green C, Bara R, Petrie Huitema CM, Ehrenkranz RA, Tyson JE, Das A, Hammond J, Peralta-Carcelen M, Evans PW, Heyne RJ, Wilson-Costello DE, Vaucher YE, Bauer CR, Dusick AM, Adams-Chapman I, Goldstein RF, Guillet R, Papile LA, Higgins RD; Eunice Kennedy Shriver NICHD Neonatal Research Network. Childhood outcomes after hypothermia for neonatal encephalopathy. N Engl J Med. 2012 May 31;366(22):2085-92. doi: 10.1056/NEJMoa1112066. PMID 22646631
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/